CLINICAL TRIAL: NCT02109510
Title: Comparative Study of Single Port Thoracoscopic Bullectomy Under Nonintubated Local and Sedation Anesthesia Versus Intubated General Anesthesia for Primary Spontaneous Pneumothorax.
Brief Title: Comparative Study of Nonintubated Anesthesia Versus Intubated General Anesthesia in Single Port Thoracoscopic Bullectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Jinwook, Hwang, Clinical Assistant Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NISIVATS01
Record Dates: First submitted 2014-03-27; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Primary Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nonintubated sedation anesthesia (Experimental): nonintubated single port thoracoscopic bullectomy using local anesthesia under sedation Drug: Dexmedetomidine IV loading dose of 1ug/kg for 10 minutes and maintain dosage of 0.3-1 ug/kg/hr, ketamine IV 2-4 mg/kg/hr and intercostal nerve block with 2% lidocaine 2cc Device: facial O2 Mask
  Interventions: Drug: nonintubated sedation anesthesia with dexmedetomidine IV, ketamine IV and intercostal nerve block with lidocaine infiltration; Procedure: single port thoracoscopic bullectomy
- Intubated general anesthesia (Active Comparator): intubated single port thoracoscopic bullectomy under general anesthesia Drug: propofol 2mg/kg IV , rocuronium 0.6mg/kg IV,1.2-2.4% sevoflurane, N20 50% 02 at fresh gas flow of 4L/min Device: double lumen endotracheal tube intubation
  Interventions: Drug: intubated general anesthesia with propofol IV, rocuronium IV ,sevoflurane and N2O gas; Procedure: single port thoracoscopic bullectomy

INTERVENTIONS:
Drug: nonintubated sedation anesthesia with dexmedetomidine IV, ketamine IV and intercostal nerve block with lidocaine infiltration
  Arms: Nonintubated sedation anesthesia
Drug: intubated general anesthesia with propofol IV, rocuronium IV ,sevoflurane and N2O gas
  Arms: Intubated general anesthesia
Procedure: single port thoracoscopic bullectomy — Thoracoscopic bullae resection with automated stapler through the single incision (2.0 cm length) at 5th intercostal space.

SUMMARY:
Investigators compared the patients' subjective postoperative symptoms and complications between the double lumen endotracheal intubated patients under general anesthesia and non-intubated patients under sedation and local anesthesia including

1. postoperative Visual scale of pain
2. postoperative sore throat/voice change
3. postoperative nausea/vomiting
4. intraoperative Arterial blood gas analysis
5. cost for anesthesia
6. morbidity

DETAILED DESCRIPTION:
Thoracoscopic bullectomy for primary spontaneous pneumothorax is relatively simple and short procedure compared to other thoracic surgery. However, in the anesthetic preparation, complicated technique and procedures are needed including a double lumen endotracheal intubation, auscultation, and flexible bronchoscopic confirmation of the tube location, even during lateral decubitus position. The double lumen endotracheal tube has a bigger outer diameter. And postoperative sore throat and voice change can develop after the intubation procedure.

Recently, single lumen intubation using carbon dioxide gas instillation under general anesthesia during thoracoscopic surgery is reported. However, if safety and efficacy are warranted, thoracoscopic surgery using nonintubated and self-ventilated anesthesia will be a best solution for above mentioned postoperative discomforts.

Investigators designed the comparative study of nonintubated local anesthesia under sedation and intubated general anesthesia in thoracoscopic bullectomy through the single port. Investigators will investigate postoperative pain, sore throat, voice change, nausea, vomiting, and intraoperative arterial blood gas analysis.

This study will be performed at Korea University Ansan Hospital. A total of 40 patients will be enrolled (20 patients in each arm).

ELIGIBILITY:
Inclusion Criteria:

1. primary spontaneous pneumothorax
2. Age between 13 and 30
3. ASA score 1,2
4. written informed consent

Exclusion Criteria:

1. A history of previous bullectomy or ipsilateral thoracic operation
2. Pregnant or lactation female
3. A cognition or mental dysfunction
4. Consumption of oral sedatives
5. A present sore throat or hoarseness
6. ASA score greater than 3

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
comparing the postoperative discomforts after intervention of each group | participants will be checked at 1 hour and 24 hours later after finishing operations
  post operative pain/sore throat/voice change

SECONDARY OUTCOMES:
intraoperative Arterial Blood Gas Analysis | during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Korea University College of Medicine, Ansan, Outside U.S and Canada, South Korea